CLINICAL TRIAL: NCT06048523
Title: Clinical and Paraclinical Characterisation of Neurogenetic Diseases, and Creation of a Hub to Facilitate Translational Research, From Basic to Clinical Research
Brief Title: Prospective Cohort Study of Neurogenetic Diseases
Acronym: CNGD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2022/73
Record Dates: First submitted 2023-06-13; First posted 2023-09-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Genetic Disease; Nervous System Diseases
Keywords: Hub; Translational research; Neurogenetics disorders; Biocollection
MeSH Terms: conditions — Genetic Diseases, Inborn; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient cohort (Other): Patients with a molecularly identified NGD (80 patients in total of which 15 with LP (Lumbar Puncture) and of which 30 with cutaneous biopsy)
  Interventions: Procedure: Patient cohort
- Control cohort (Other): Patients control: 10 controls with lumbar puncture and 10 controls without LP (Lumbar Puncture)
  Interventions: Procedure: Control cohort

INTERVENTIONS:
Procedure: Patient cohort — * For patients: annual follow-up in Neurogenetic reference center, as part of routine care, with exhaustive standardised clinical evaluation
  * Paraclinical monitoring (e.g. MRI, EEG, EMG, etc.) modelled on standard care according to current recommendations
  * Biological samples offered to patients in the context of research:
    * Annual blood sample
    * Annual urine sample
    * Collection of 1 skin biopsy at the inclusion visit (for 30 patients)
    * Cerebrospinal fluid sample at the inclusion visit (for 15 patients
  Arms: Patient cohort
Procedure: Control cohort — * controls without LP: 1 visit for blood, urine and optional skin biopsy
  * controls with LP: additional blood and cerebrospinal fluid tubes for blood sampling and LP as part of routine care, without longitudinal follow-up
  Arms: Control cohort

SUMMARY:
Neurogenetic diseases (NGD) represent rare and hereditary forms of neurological diseases. The goal of CNGD is to create a one-window approach for NGDs, to facilitate and accelerate participation in research projects through deep phenotyping and the availability of low-cost biological samples for research teams. It is positioned as a true hub allowing new connections between clinical and basic research teams and ultimately as an incubator for translational projects for NGDs, in order to be able to initiate therapeutic trials, the ultimate objective of clinical and translational research.

DETAILED DESCRIPTION:
Neurogenetic diseases (NGDs) represent rare inherited forms of neurological diseases. They constitute a constellation of different diseases, affecting neurodevelopment (syndromic or non-syndromic intellectual disabilities (ID), with or without autism spectrum disorders (ASD), epileptic encephalopathies, neurodevelopmental disorders (NDD) with or without ID... ) or leading to early neurodegeneration (Huntington's and Huntington-like disease, hereditary ataxias, hereditary spastic paraplegias (HSP), primary dystonias, neurodegeneration due to intracerebral iron accumulation (NBIA), neurometabolic diseases, etc.). Progress in the knowledge of the genetic causes of NGDs is unceasing, with the discovery of new genes involved in their determinism being continuous. As a result, the boundary between routine care and clinical research is extremely narrow and blurred, and the two activities are totally intertwined and interdependent in the care of patients.

For patients with NGDs already characterized by molecular genetics, at an early, intermediate or presymptomatic stage, we will perform a comprehensive annual standardized clinical and paraclinical evaluation for deep phenotyping as part of routine care; collection of biological samples (annual blood and urine sampling, optional skin biopsy and optional cerebrospinal fluid (CSF) sampling), for functional analyses and better understanding of the pathophysiological mechanisms involved. This study will last 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patient-specific inclusion criteria
* Age ≥ 6 years
* Patient with a molecularly identified NGD

  o Specific inclusion criteria for controls
* For the 10 controls with lumbar puncture (LP): person who performed an LP for medical reasons and who consented to participate in the collection of biological samples
* Age ≥ 18 years
* Person matched in age (+/- 5 years) and sex to adult patient with NGD at the time of collection

Exclusion Criteria:

* Participation in an interventional clinical trial that may interfere with our study
* Refusal of blood collection
* Pregnant and breastfeeding women
* Only for patients performing LP: Contraindication to LP
* Specific non-inclusion criteria for controls: Criterion of a neurodegenerative or inflammatory pathology of the central nervous system

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Constitution of a biobank of NGD patients correlated with clinical data | Inclusion visit, 12 months visit and 24 months visit
  Number of participants for whom minimum clinical data have been collected and for whom at least one at least one protocol sample has been collected

CONTACTS AND LOCATIONS:
Overall Officials: Chloe ANGELINI, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Bordeaux, France